CLINICAL TRIAL: NCT04022434
Title: Investigation of Supplemental L-alanine in the Management of Dietary Fructose Intolerance: a Double-blind, Randomized Study
Brief Title: Investigation of Supplemental L-alanine in the Management of Dietary Fructose Intolerance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 611777
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-07

CONDITIONS: Fructose Intolerance
MeSH Terms: conditions — Fructose Intolerance | interventions — Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Psyllium powder is used as the placebo. A member of the research staff will package and dispense L-alanine and placebo in similar containers. A standard measuring spoon will be provided to the subject for preparing the placebo solution. Subjects will mix the placebo in the beverage of their choice and consume this approximately 20 minutes before meals or snacks, in according with the dosing guidelines set for them by the dietitian.
  Meal Placebo Breakfast * 1-2 scoops Snack * .5 - 1 scoop Lunch * 1-2 scoops Snack * .5 - 1 scoop Dinner * 1-2 scoops
  Interventions: Dietary Supplement: Placedo
- Experimental Alanine (Experimental): L-alanine, USP (Spectrum® Chemicals and Laboratory Products, Gardena, CA) will be packaged and dispensed by one member of the research staff who will have no other role in the study. A one-month supply will be dispensed to the subjects.
  Meal L-Alanine Breakfast * 1-2 scoops Snack * .5 - 1 scoop Lunch * 1-2 scoops Snack * .5 - 1 scoop Dinner * 1-2 scoops
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Placedo — Subjects will mix the placebo in the beverage of their choice and consume this approximately 20 minutes before meals or snacks, in according with the dosing guidelines set for them by the dietitian.
  Arms: Placebo
Dietary Supplement: Alanine — Subjects will mix the alanine in the beverage of their choice and consume this approximately 20 minutes before meals or snacks, in according with the dosing guidelines set for them by the dietitian.
  Arms: Experimental Alanine

SUMMARY:
Over the past few decades, fructose consumption has risen significantly in the United States1. This sugar is increasingly being used as a sweetener in a variety of foods1. Because there is a limited absorptive capacity for fructose, excessive ingestion of fructose leads to fructose malabsorption and dietary fructose intolerance (DFI) 2-9, 13. Incomplete absorption of fructose may lead to a variety of gastrointestinal symptoms, including bloating, pain, gas and diarrhea 2-9. In tertiary care centers, the prevalence of DFI in subjects with unexplained GI symptoms has been estimated to range between 11-50 %, when subjects were assessed with breath tests following administration of 25 grams of fructose 2, 5-7.

Currently, the main treatment for DFI consists of restricting the intake of fructose-containing foods 10-12 or limiting the intake of foods with excess "free fructose" (ie, fructose in excess of glucose) or a high fructan content17. These diet restrictions can improve symptoms in patients with DFI 10-12,17. However, the diet is very restrictive and imposes a significant burden on the individual and the family. In one study, 40% of subjects were unable to comply with dietary restrictions 10. Currently, there are no other therapeutic agents for treating this condition 14, 15. Apart from promoting intestinal fructose absorption, an ideal therapeutic agent should be safe, simple to use, inexpensive and have no calorific value.

Fructose is mostly absorbed in the small intestine by facilitated diffusion which is mediated by the GLUT-5 transporter protein. This protein is expressed on the intestinal mucosal surface. In the presence of glucose, fructose absorption is increased, mostly due to co-transport with glucose via the GLUT-2 transporter protein. However, the calorie content of glucose precludes its routine use in patients with DFI. Other compounds that promote fructose absorption, such as 3 O-methyl glucose and epidermal growth factor (EGF) have significant side effects and safety issues, making them unsuitable for clinical use in DFI.

Several amino acids, including alanine, have been also been shown to increase intestinal fructose absorption 14. The postulated mechanism is as follows: transmucosal Na+-coupled amino acid transport causes increased water flow through the mucosal apical membrane14. This, in turn, facilitates fructose absorption by a process of 'solvent drag', caused by an increase in intraluminal fructose concentration caused by water removal from the lumen14. The potential benefit of alanine was assessed in a European study in healthy children 14. Ten subjects underwent H2 breath tests following administration of fructose alone (2g/ Kg body weight), followed by a combination of fructose and an equi-molar dose of various amino acids (L-alanine, L-phenylalanine, L-glutamine, L-proline) or glucose. Breath H2 production was assessed as a marker of intestinal fructose absorption. Subjects were asked to report any gastrointestinal symptoms during the test. All subjects had a positive (>20 ppm of H2) breath test (68 ± 38 ppm) with fructose and 6/10 subjects reported either abdominal pain or diarrhea during the test. Co-administration of alanine caused a significant (p < 0.05) decrease in breath H2 production (3 ± 3 ppm), suggesting increased intestinal fructose absorption. Furthermore, none of the subjects reported any gastrointestinal symptoms during the test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fructose malabsorption (positive breath test after ingestion of 25 grams of fructose defined as either (a) ≥ 20 ppm rise of breath H2/CH4/both over baseline values or a successive rise of ≥ 5 ppm over baseline and in 3 consecutive breath samples)
* Women of childbearing potential must agree to a urine pregnancy test before supplement is dispensed and to avoid pregnancy throughout the study.

Exclusion Criteria:

* Cognitive impairment or any other inability to provide informed consent
* Prisoners
* GI surgery except appendectomy, cholecystectomy, caesarean section, hysterectomy
* Antibiotics in the previous 6 weeks.
* Major co-morbid illnesses, including chronic pancreatitis, celiac disease, inflammatory bowel disease, diabetes, scleroderma, pseudo-obstruction syndromes etc.
* Medication use: opioids, Tegaserod, laxatives, enemas
* Difficulty Swallowing
* Known food allergies or intolerance to any fiber supplements or other dietary nutritional supplements such as: Psyllium (Metamucil), Maltodextrin, Citric Acid, and methylcellulose (Citrucel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2014-01-07 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
GI symptom score | 4 weeks
  Change in GI symptom score with alanine and placebo, when compared to the baseline

SECONDARY OUTCOMES:
Fructose consumption | 4 weeks
  Estimated daily consumption of fructose during the alanine and placebo phases, when compared to the baseline using prospective food diaries
Breath hydrogen and methane | 4 weeks
  Changes in breath hydrogen and/or methane values with alanine and placebo when compared with to the baseline
Quality of Life (SF-12) | 4 weeks
  Changes in SF-12 scores between and after baseline and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States